CLINICAL TRIAL: NCT00668421
Title: A Multicenter, Open Label Phase I/II Study of CEP-701 (Lestaurtinib) in Adults With Myelofibrosis
Brief Title: CEP-701 (Lestaurtinib) in Myelofibrosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ronald Hoffman (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ronald Hoffman, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 07-0548-00104; P01CA108671-01A2 (NIH); MPD-RC 104 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Myelofibrosis; Essential Thrombocythemia; Polycythemia Vera
Keywords: Myelofibrosis; Essential Thrombocythemia; Polycythemia Vera; JAK2 V617F Mutation; Lestaurtinib
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera | interventions — lestaurtinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CEP-701 (Lestaurtinib) (Experimental): Subject is to receives Lestaurtinib, in Phase 1: standard cohort dose escalation; Phase 2: single stage design to estimate the percentage of subjects with a 15% or greater reduction in JAK2 V617F allele frequency in peripheral blood granulocytes in 6 months of treatment
  Interventions: Drug: CEP-701 (Lestaurtinib)

INTERVENTIONS:
Drug: CEP-701 (Lestaurtinib) — Lestaurtinib (CEP-701), oral formulation. Phase 1: 80 BID - 160 BID; phase 2: 140 mg

SUMMARY:
Myelofibrosis is the gradual replacement of bone marrow (place where most new blood cells are produced) by fibrous tissue which reduces the body's ability to produce new blood cells and results in the development of chronic anemia (low red blood cell count). One of the main distinctions of myelofibrosis is "extramedullary hematopoesis", the migration or traveling of the blood-forming cells out of the bones to other parts of the body, such as the liver or spleen, resulting in an enlarged spleen and liver.

Treatment for myelofibrosis is unsatisfactory and there is no medication that is specifically used in the treatment of myelofibrosis. There is a protein that is found to be present in the majority of myelofibrosis patients (JAK2) and the drug Lestaurtinib is being studied to see if it will stop this protein from functioning and thereby help control the disease.

This study is divided into two Phases (1 & 2). In phase 1 we will be looking for the dose of study medication (Lestaurtinib) that will be the highest dose a patient can take without experiencing serious side effects, maximum tolerated dose (MTD).

In phase 2, after the MTD dose has been established in phase 1, we will be investigating how well CEP-701 (Lestaurtinib) works at suppressing the protein (JAK2).

The investigators also wish to find out important biologic characteristics or features of myelofibrosis through an additional correlative biomarker study (MPD-RC #107). The correlative biomarker study is a study that is related to the main study, but is looking to answer different questions than the main study. The purpose of the biomarker study is to understand the causes of MPD and to develop improved methods for the diagnosis and treatment of these diseases, while the main study is trying to find out how well CEP-701 (Lestaurtinib) will work in treating the myeloproliferative disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary myelofibrosis, essential thrombocythemia related myelofibrosis, or polycythemia vera related myelofibrosis requiring therapy, including:

   1. those previously treated and relapsed or refractory
   2. or newly diagnosed, with intermediate or high risk according to Lille Scoring system (adverse prognostic factors are: Hb < 10 g/dl, WBC < 4 or > 30 x 109/L; risk group: 0 = low, 1 = intermediate, 2 = high)
   3. or with symptomatic splenomegaly (must be >=10 cm below the left costal margin in the mid-clavicular line).
2. The subject must not be considered as a candidate to receive allogeneic hematopoietic stem cell transplant at the time of being enrolled into the study.
3. The subject has a detectable JAK2 V617F mutation.
4. Signed informed consent: Patients must have signed consents for both the Lestaurtinib protocol and for the mandatory biomarker MDP-RC 107 protocol to be eligible to participate.
5. Patients must have been off any PMF-directed therapy for 4 weeks prior to entering this study and have recovered from the toxic effects (grade 0-1) of that therapy. Treatment with erythropoietin is permitted.
6. Serum bilirubin levels less than or equal to 2 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed by treating physician to active hemolysis or ineffective erythropoiesis due to myelofibrosis.
7. Serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels less than or equal to 2 x ULN.
8. Serum creatinine levels less than or equal to 1.5 x ULN.
9. Women of childbearing potential must have a negative serum or urine pregnancy test prior to Lestaurtinib treatment and should be advised to avoid becoming pregnant. Men must be advised to not father a child while receiving treatment with Lestaurtinib. Both women of childbearing potential and men must practice effective methods of contraception (those generally accepted as standard of care measures). Women of child bearing potential are women who are not menopausal for 12 months or who have not undergone previous surgical sterilization. If the subject is a woman of childbearing potential, she must use a medically acceptable form of contraception during the study period and for 30 days thereafter. If the subject is a man he must be surgically sterile or must use a medically approved method of contraception for the duration of the study and for 60 days following the last dose of CEP-701.
10. Age > 18 years.

Exclusion Criteria:

1. Nursing and pregnant females. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
3. Unstable angina.
4. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days, or anticipation of the need for major surgical procedure during the course of the study.
5. Biopsy or other minor surgical procedure, excluding placement of a vascular access device or bone marrow biopsy, within 7 days prior to study enrollment.
6. Ongoing serious, non-healing wound, ulcer, or bone fracture.
7. Known hypersensitivity to any component of Lestaurtinib.
8. The subject has received a donor stem cell transplant in the past and has detectable full or partial donor chimerism.
9. The subject requires treatment with a CYP3A4 inhibitor, including azole antifungals (topicals are permitted); protease inhibitors; nefazodone; cyclosporine; erythromycin; clarithromycin; and troleandomycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2013-09 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and maximum tolerated dose of a novel kinase inhibitor in subjects with myelofibrosis. | 2 years
To estimate the efficacy of a novel kinase inhibitor in subjects with myelofibrosis, as determined by a reduction in JAK2 V617F allele frequency in peripheral blood neutrophils. | 2 years

SECONDARY OUTCOMES:
To estimate the incidence, severity, and attribution of treatment-emergent adverse events. | 2 years
To estimate the rate of complete or major clinical-hematological response from treatment with Lestaurtinib (CEP-701) in this subject population as measured by the EUMNET response criteria. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hoffman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (7):
- United States (7):
  - Palo Alto Medical Facilities, Palo Alto, California
  - Georgetown University Medicine Center, Washington D.C., District of Columbia
  - University of Maryland Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Weill Cornell, Ithaca, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Hexner EO, Mascarenhas J, Prchal J, Roboz GJ, Baer MR, Ritchie EK, Leibowitz D, Demakos EP, Miller C, Siuty J, Kleczko J, Price L, Jeschke G, Weinberg R, Basu T, Pahl HL, Orazi A, Najfeld V, Marchioli R, Goldberg JD, Silverman LR, Hoffman R. Phase I dose escalation study of lestaurtinib in patients with myelofibrosis. Leuk Lymphoma. 2015;56(9):2543-51. doi: 10.3109/10428194.2014.1001986. Epub 2015 Feb 20. PMID 25563429